CLINICAL TRIAL: NCT00356239
Title: Evaluation of Safety and Feasibility Magnetic Resonance Imaging of the Heart at 1.5 Tesla In Patients With Implantable Cardioverter Defibrillators
Brief Title: Implantable Cardioverter Defibrillators And Magnetic Resonance Imaging of the Heart at 1.5 Tesla
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Bonn (Other)
Other Study IDs: 201/05
Record Dates: First submitted 2006-07-24; First posted 2006-07-25 (Estimated); Last update posted 2007-04-11 (Estimated); Status verified 2007-04

CONDITIONS: Defibrillators, Implantable; Heart Failure, Congestive
Keywords: Defibrillators, Implantable; Heart Failure, Congestive; Magnetic Resonance Imaging
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Observational Model: Defined Population | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
To evaluate short-term and long-term effects by MR imaging on the technical and functional status of implantable cardioverter defibrillators.

DETAILED DESCRIPTION:
The presence of an implantable cardioverter defibrillators (ICD) is currently considered an absolute contraindication to MR imaging, and most patients with PM are excluded from having MRI. As a result from studies such as MADIT I, MADIT II, SCDHeft etc. the number of patients with ICDs has been continuously growing over the past years, ans this development will continue.

The aim of this study is to develop a strategy for safe performance of MR imaging at 1.5T, which included restriction of specific absorption rate (SAR) values to minimize the risk of lead heating, and ICD reprogramming to avoid interference from time varying gradient fields. The safety of this approach is then evaluated in a large group of ICD patients including assessment of potential myocardial thermal injury by measuring serum troponin I and pacing capture thresholds, and performing a follow-up 6 weeks after MR imaging to evaluate long-term effects.

ELIGIBILITY:
Inclusion Criteria:

* Implantable Cardioverter Defibrillator
* congestive heart failure
* informed consent

Exclusion Criteria:

* Non-MRI-compatible implants

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 25
Dates: Start 2006-07

CONTACTS AND LOCATIONS:
Overall Officials: Nikos Werner, MD, Principal Investigator — University of Bonn, Department of Cardiology
Locations (1):
- University of Bonn, Department of Cardiology, Bonn, North Rhine-Westphalia, Germany

REFERENCES:
- [Derived] Naehle CP, Strach K, Thomas D, Meyer C, Linhart M, Bitaraf S, Litt H, Schwab JO, Schild H, Sommer T. Magnetic resonance imaging at 1.5-T in patients with implantable cardioverter-defibrillators. J Am Coll Cardiol. 2009 Aug 4;54(6):549-55. doi: 10.1016/j.jacc.2009.04.050. PMID 19643318